CLINICAL TRIAL: NCT03078764
Title: The Adaptation, Usability, and Feasibility of a Mobile Health (mHealth) System to Improve Type 2 Diabetes Self-management in Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Mahidol University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Panan Pichayapinyo, Associate Professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00118973; 5D43TW009883-03 (NIH)
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Mobile health (mHealth)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Arm using mHealth (Experimental): Patients with uncontrolled type 2 diabetes
  Interventions: Other: Mobile health system
- Community nurses (Experimental): Nurses who receive mHealth report about patients in the patients' arm.
  Interventions: Other: E-mail reports and technical support for mHealth system

INTERVENTIONS:
Other: Mobile health system — Patients will receive weekly automated IVR telephone calls for 12 weeks to assess their glycemic symptoms, medication adherence, dietary consumption, physical activity, sleep, and foot care. These 5-10 minute calls will follow a standardized Thai language IVR script developed specifically for this study.
  Other Names: mHealth; Interactive Voice Response (IVR)
  Arms: Patient Arm using mHealth
Other: E-mail reports and technical support for mHealth system — Nurses will also receive a technical troubleshooting guide, and have similar access to live telephone technical support. Once their patients' calls begin, nurses will begin receiving weekly e-mail reports summarizing each patients' assessment results, any active self-management problems the patients reported, and suggested strategies for supporting the patient's self-management.
  Arms: Community nurses

SUMMARY:
This project explores the feasibility of using automated telephone calls to adult patients with type 2 diabetes to improve diabetes self-management in Thailand. This line of work could significantly extend Thai nurses' ability to manage this growing epidemic, and ultimately reduce the suffering and costs caused by diabetes in Thailand.

DETAILED DESCRIPTION:
There is a serious shortage of community nurses to address Thailand's significant and expanding burden of poorly controlled type 2 diabetes. However, mobile health (mHealth) strategies are likely to significantly improve and extend Thai nurses' ability to monitor and manage these patients. This study aims to:

1) investigate the feasibility and acceptability of a culturally- and clinically-adapted mHealth intervention with adult Thai diabetic patients and their community nurses, and 2) estimate the intervention's effect upon glycated hemoglobin (HbA1c), fasting blood glucose, self-management behaviors, and diabetes-related distress in uncontrolled type 2 diabetes. Thirty-six patients with poorly controlled type 2 diabetes (along with their regular nurses) will be recruited through an established community clinic network. After baseline clinical and behavioral assessment, patients will receive 12 weeks of automated 10-minute weekly Interactive Voice Response (IVR) calls to provide monitoring and self-management support related to glycemic symptoms, medication adherence, and several self-care behaviors. Patients' clinical nurse will receive weekly summaries of each IVR call by text message and email with guidance on Thai-appropriate best practices. Principal investigator will receive email whenever patients report a potentially urgent issue by IVR, i.e., symptoms of hypoglycemia, or inadequate supply of medication. Immediately after the 12-week intervention concludes, clinical and behavioral variables will be reassessed and a mixed-methods process evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

For patients:

1. poorly controlled type 2 diabetes as indicated by HbA1c ≥ 7.5% recorded within past 6 months
2. aged 20 years and older
3. currently being treated by oral antihyperglycemic
4. communicates and reads in Thai
5. has access to and able to use a touch-tone phone (either a land line or a mobile phone)
6. free of major physical, cognitive, or psychiatric impairment (per medical records and PI discretion) that would prevent them from participating meaningfully in the intervention.

Inclusion criteria:

For nurses:

1. works in a non-communicable disease clinic.
2. can access email
3. has a mobile telephone.

Exclusion Criteria:

For patients:

1. have participated in other mHealth interventions within 3 months
2. have baseline HbA1c < 7.5%
3. are hospitalized or otherwise at risk for hospitalization
4. are prescribed injected insulin
5. patients and nurses who participated in the usability trial will be ineligible to participate in the pilot trial.

Exclusion criteria:

For nurses: None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 13 weeks
  It refers to glycated haemoglobin, which identifies average plasma glucose concentration.
Diabetes related distress | 13 weeks
  It will be measured using the emotional and regimen subscales of a Thai translation of the well-validated Diabetes Distress Scale. This is a reliable and validated scale, and correlates with other measures of emotional distress. The responses range from 1-6. The higher scores indicate a greater degree of distress.

SECONDARY OUTCOMES:
Fasting blood glucose | 13 weeks
  It refers to blood glucose levels after refraining eating or drinking for at least 8 hours.

OTHER OUTCOMES:
Sleep quality | 13 weeks
  It will be assessed using the same single item used during the IVR assessment, along with the PROMIS Sleep Disturbance-Short Form. The PROMIS (Patient-Report Outcomes Information System) Sleep Disturbance-Short Form is a 4-item self-report instrument covering the quality of sleep-wake functioning. Responses are scored on a 5-point Likert scale. The higher scores indicating a greater degree of sleep disturbance.
Dietary consumption | 13 weeks
  It will be assessed using the same single item used during the IVR assessment. The responses range from 0 to 7 (days).
Physical activity | 13 weeks
  It will be assessed using the Stanford Leisure-Time Activity Categorical Item (Kiernan et al., 2013), which consists of 6 descriptive categories ranging from inactive (1) to very active, almost daily physical activity (6).
Foot care | 13 weeks
  It will be assessed using the same single item used during the IVR assessment. The responses range from 0 to 7 (days).
Symptoms of hypoglycemia | 13 weeks
  It will be assessed using a 7 items that ask about low blood sugar symptoms, the same that the study team describe in the IVR calls. The responses range from 0 (not at all) to 4 (6-7 days a week). The higher scores indicate a greater degree of hypoglycemic symptoms.
Depressive symptoms severity | 13 weeks
  It will be assessed using the Patient Health Questionnaire-8 (PHQ-8) (Kroenke et al., 2009). It consists of 8 items with a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). Higher scores indicate greater depressive symptom severity.
Readiness for change | 13 weeks
  It will be assessed using 5 items from our prior research that is specifically worded to measure participants'preparedness to change the 5 diabetes self-care behaviors that our program targets, which are answered using a 7-point Likert scale ranging from 1 (not at all) to 7 (very much so). Higher scores indicate greater readiness for change.
Diabetes self-efficacy | 13 weeks
  It will be assessed with the Self-Efficacy for Diabetes Scale (Ritter et al., 2016). The scale consists of 8 items with 10- point Likert scale ranging from 1 (not at all confident) to 10 (totally confident). Higher scores indicate greater self-efficacy.
Medical adherence | 13 weeks
  It will be assessed using the Hill-Bone Compliance Scale (Kim et al., 2000), assesses how often patients miss taking medications, rated on a 4-point Likert scale ranging from 1(none of the time) to 4 (all of the time). In the study, only 8 items of Hill-Bone Compliance scale will be used. Reverse coded before analysis will be performed. Higher scores indicate greater medication adherence. In addition, 1-item of the Brief Medication Questionnaire will be used, which allows calculation of percent adherence over the past 2 weeks
Social support | 13 weeks
  It will be assessed using selected items from the Norbeck Social Support Questionnaire, which is a validated measure of number, type, and quality of relationships (Norbeck, 1983). For the purpose of this study, the 6 items (item 3-8) will be scored on a 5-point Likert scale ranging from 0 (not at all) to 4 (a great deal). Higher scores indicate better social support.
Health literacy | 13 weeks
  It will be assessed using the 3-item screener developed by Chew et al. for detecting probable inadequate health literacy (45, 46). Higher scores indicate better health literacy.
Client satisfaction | 13 weeks
  will be measured using the Client Satisfaction Questionnaire (CSQ-8) (Attkisson, Zwick, 1982), which assesses satisfaction with specific providers, settings, and time intervals, along with open-ended items (within the exit interview) adapted from prior mHealth research studies. Higher scores indicate greater satisfaction of the program.
Self-efficacy (for nurse) | 13 weeks
  It will be measured using Nurse Self-efficacy for Diabetes Care using 11 items developed for this study that correspond to patients' IVR content areas.

CONTACTS AND LOCATIONS:
Overall Officials: Panan Pichayapinyo, PhD., Principal Investigator — University of Michigan
Locations (6):
- Thailand (6):
  - Buengbon Health Promoting Hospital, Nong Suea, Changwat Pathum Thani
  - Buengkasam 1 Health Promoting Hospital, Nong Suea, Changwat Pathum Thani
  - Buengkasam 2 Health Promoting Hospital, Nong Suea, Changwat Pathum Thani
  - Buengshamaor 1 Health Promoting Hospital, Nong Suea, Changwat Pathum Thani
  - Nongsamwang 1 Health Promoting Hospital, Nong Suea, Changwat Pathum Thani
  - Salakru Health Promoting Hospital, Nong Suea, Changwat Pathum Thani

IPD SHARING:
Plan to Share IPD: No